CLINICAL TRIAL: NCT06846593
Title: The Comparison and Combination of Semiconductor Embedded Therapeutic Arm Sleeves and Platelet-Rich Plasma With Adipose Stem Cell (PRP+ASC) Injections for the Treatment of ECRB Tendinopathy (Lateral Epicondylitis): A Randomized, Double-Blinded, Placebo-Controlled Prospective Clinical Trial
Brief Title: The Comparison of Semiconductor Embedded Therapeutic Arm Sleeves for the Treatment of ECRB Tendinopathy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCG IRB Protocol #20242832; 2024-06 (Other: Incrediwear)
Record Dates: First submitted 2024-11-13; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: ECRB Tendinopathy
Keywords: ECRB; lateral epicondylitis; tendinopathy; tennis elbow; extensor carpi radialis brevis; platelet-rich plasma; PRP; stem cell therapy; arm sleeves
MeSH Terms: conditions — Tennis Elbow; Tendinopathy | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Subjects will determine whether they would like to receive Standard of Care (SOC) PRP+ASC injections. Then, the subjects will be randomly assigned to the study group in which they will receive a real or sham semiconductor embedded sleeve. The subjects will be instructed to wear the sleeve for a minimum of 12 hours per day, including overnight, for the entire duration of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Incrediwear only (Active Comparator): One group will receive active therapy (semiconductor embedded arm sleeve) "Incrediwear only"
  Interventions: Device: Semiconductor Embedded Therapeutic Arm Sleeves
- Sham Incrediwear (Sham Comparator): One group will receive placebo therapy (arm sleeve absent of semiconductor thread) "Sham Incrediwear"
  Interventions: Device: Placebo Arm Sleeves
- Incrediwear with PRP+ASC injections (Active Comparator): One group will receive active therapy with SOC (standard of care) PRP+ASC injections (active semiconductor embedded arm sleeves after they have received PRP+ ASC injections as part of their routine care) "Incrediwear with SOC PRP+ASC injections"
  Interventions: Device: Semiconductor Embedded Therapeutic Arm Sleeves; Other: Platelet-Rich Plasma with Adipose Stem Cell (PRP+ASC) Injections
- Sham Incrediwear with PRP+ASC injections (Sham Comparator): One group will receive placebo therapy with SOC (standard of care) PRP+ASC injections (arm sleeve absent of semiconductor fabric after they have received PRP+ASC injections as part of their routine care) "Sham Incrediwear with SOC PRP+ASC injections"
  Interventions: Device: Placebo Arm Sleeves; Other: Platelet-Rich Plasma with Adipose Stem Cell (PRP+ASC) Injections

INTERVENTIONS:
Device: Semiconductor Embedded Therapeutic Arm Sleeves — labeled A or B, assigned based on blinded randomization table provided by the sponsor.
  Arms: Incrediwear only; Incrediwear with PRP+ASC injections
Device: Placebo Arm Sleeves — labeled A or B, assigned based on blinded randomization table provided by the sponsor.
  Arms: Sham Incrediwear; Sham Incrediwear with PRP+ASC injections
Other: Platelet-Rich Plasma with Adipose Stem Cell (PRP+ASC) Injections — patients will choose or opt out of these standard of care injections.
  Arms: Incrediwear with PRP+ASC injections; Sham Incrediwear with PRP+ASC injections

SUMMARY:
This study seeks to identify patient reported and clinically measured outcomes for pain management and elbow function with application of semiconductor embedded fabric combined with PRP+ASC injections in the affected area.

DETAILED DESCRIPTION:
Extensor Carpi Radialis Brevis (ECRB) tendinopathy, also known as lateral epicondylitis or tennis elbow, is the most prevalent elbow soft tissue injury and affects 1-3% of the population. Repetitive overloading of the tendon and ligaments in the elbow lead to microtraumas, causing abnormal angiofibroblastic remodeling and increased pain. Microtearing occurs most commonly at the origin of the extensor carpi radialis brevis (ECRB) tendon. The main symptoms include a loss of grip strength, a burning sensation near the ECRB origin site, and pain during daily activities such as grasping objects or shaking hands. Both conditions present a significant injury and treatment burden on the population and effective treatment and pain management approaches with minimal side effects are needed.

Novel nonsurgical treatment approaches for ECRB tendinopathy include platelet-rich plasma (PRP) injections and stem cell therapy. Ultrasound-guided PRP and adipose-derived stem cells (ASCs) injections have shown to be an effective treatment option for patients with chronic ECRB tendinopathy.

The proposed study seeks to assess the effect of non-compressive semiconductor embedded arm sleeves in combination with PRP + ASC injections, throughout a 6-month rehabilitation course for patients with ECRB tendinopathy. Outcome measures will be collected at standardized intervals to evaluate and compare treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ECRB tendinopathy as determined by radiographic assessment or ultrasound imaging.
2. Patients age 18-65
3. Patients who are willing and able to adhere to follow-up schedule and protocol guidelines.
4. Patients who are willing and able to sign corresponding research subject consent form.

Exclusion Criteria:

1. Patient has a history of neurological conditions, including multiple sclerosis or Parkinson's disease
2. Patient has severe medical condition, including recent myocardial infarction, unstable angina, heart failure, severe anemia
3. Patient has had prior surgical treatment of the elbow in the last 5 years or injection treatment(s) in the last 2 years
4. Patient has complete tear of ECRB tendon or other surgical indication
5. Patient has chronic pain conditions unrelated to elbow condition
6. Patient has auto-immune or auto-inflammatory diseases
7. Patient has used tobacco within the last 90 days
8. Patient is not within the ages of 18-65
9. Patient has a history of metabolic disorders
10. Patient has an active infection (local or systemic)
11. Patient is unwilling or unable to sign the corresponding research subject consent form
12. Patient meets any other criteria or has any other condition that, in the opinion of the investigator, would prevent them from completing the study or that, in the opinion of the investigator, would confound study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-16 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in patient elbow function and pain as determined by the Patient-Rated Tennis Elbow Evaluation (PRTEE). | 6 months
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is a self-administered questionnaire that assesses elbow pain and functional ability in patients with tennis elbow. The minimum number is zero meaning no pain and the maximum number is 10 meaning the worst imaginable pain. Lower scores are ideal while higher scores are indicative of the patient in a lot of pain and minimal functional ability

SECONDARY OUTCOMES:
Change in pain as determined by the Visual Analog Scale (VAS). | 6 months
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The minimum number is zero meaning no pain and maximum number is 10 meaning the most pain the patient has every felt in their entire life. Lower scores are ideal while higher scores are indicative of the patient in a lot of pain.
Change in patient elbow function as determined by the Disabilities of the Arm, Shoulder, and Hand (DASH). | 6 months
  The Disabilities of the Arm, Shoulder, and Hand (DASH) is a self-administered questionnaire that assesses the patient's functional ability and arm, shoulder, or hand pain. It is on a 5-point likert scale with 1= No difficulty, 2 = Mild difficulty, 3 = Moderate difficulty, 4 = Severe difficulty, and 5 = Unable. The score ranges from 0 to 100, with higher scores indicating greater disability.
Change in grip strength as measured by a hand dynamometer | 6 months
  Patient's grip strength will be assessed with a hand dynamometer. The patient will squeeze the device with the patient's elbow at 90 degrees of flexion and wrist in 30 degrees of extension. A force output value in pounds (lbs) will be displayed and a higher number of force output indicates a stronger grip strength.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Matthew Bayes, MD, Medical, Principal Investigator — Bluetail Medical Group
Locations (1):
- Bluetail Medical Group, Chesterfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data will be stored and used for the duration of time required to conduct analysis and publish all proposed peer-reviewed papers, according to study objectives. Data will be retained for 2 years after publication to allow for re-analysis that may be initiated in response to readers/reviewers. Subject records will be maintained at the PI's clinical site for a minimum of 7 years following latest study follow-up.

REFERENCES:
- [Background] Bisset LM, Collins NJ, Offord SS. Immediate effects of 2 types of braces on pain and grip strength in people with lateral epicondylalgia: a randomized controlled trial. J Orthop Sports Phys Ther. 2014 Feb;44(2):120-8. doi: 10.2519/jospt.2014.4744. Epub 2014 Jan 9. PMID 24405258
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Rompe JD, Overend TJ, MacDermid JC. Validation of the Patient-rated Tennis Elbow Evaluation Questionnaire. J Hand Ther. 2007 Jan-Mar;20(1):3-10; quiz 11. doi: 10.1197/j.jht.2006.10.003. PMID 17254903
- [Background] Beaton DE, Katz JN, Fossel AH, Wright JG, Tarasuk V, Bombardier C. Measuring the whole or the parts? Validity, reliability, and responsiveness of the Disabilities of the Arm, Shoulder and Hand outcome measure in different regions of the upper extremity. J Hand Ther. 2001 Apr-Jun;14(2):128-46. PMID 11382253
- [Background] Cho SY, Roh YS, Roh HT. Evaluation of tympanic temperature and thermal sensation responses during exercise to verify the positive effects of wearing germanium-coated functional clothing. J Phys Ther Sci. 2016 Jun;28(6):1860-3. doi: 10.1589/jpts.28.1860. Epub 2016 Jun 28. PMID 27390434
- [Background] Kyselovic J, Masarik J, Kechemir H, Koscova E, Turudic II, Hamblin MR. Physical properties and biological effects of ceramic materials emitting infrared radiation for pain, muscular activity, and musculoskeletal conditions. Photodermatol Photoimmunol Photomed. 2023 Jan;39(1):3-15. doi: 10.1111/phpp.12799. Epub 2022 May 21. PMID 35510621
- [Background] Park JH, Lee S, Cho DH, Park YM, Kang DH, Jo I. Far-infrared radiation acutely increases nitric oxide production by increasing Ca(2+) mobilization and Ca(2+)/calmodulin-dependent protein kinase II-mediated phosphorylation of endothelial nitric oxide synthase at serine 1179. Biochem Biophys Res Commun. 2013 Jul 12;436(4):601-6. doi: 10.1016/j.bbrc.2013.06.003. Epub 2013 Jun 10. PMID 23756809
- [Background] Leung TK. In Vitro and In Vivo Studies of the Biological Effects of Bioceramic (a Material of Emitting High Performance Far-Infrared Ray) Irradiation. Chin J Physiol. 2015 Jun 30;58(3):147-55. doi: 10.4077/CJP.2015.BAD294. PMID 26014120
- [Background] Duranti C, Bagni G, Iorio J, Colasurdo R, Devescovi V, Arcangeli A. Effects of Germanium embedded fabric on the chondrogenic differentiation of adipose derived stem cells. Tissue Cell. 2024 Oct;90:102507. doi: 10.1016/j.tice.2024.102507. Epub 2024 Jul 30. PMID 39128191
- [Background] Justice TE, Jacob PB. Non-compressive sleeves versus compression stockings after total knee arthroplasty: A prospective pilot study. J Orthop. 2023 Nov 24;49:102-106. doi: 10.1016/j.jor.2023.11.044. eCollection 2024 Mar. PMID 38094981
- [Background] Vatansever F, Hamblin MR. Far infrared radiation (FIR): its biological effects and medical applications. Photonics Lasers Med. 2012 Nov 1;4:255-266. doi: 10.1515/plm-2012-0034. PMID 23833705
- [Background] Marino K, Lee R, Lee P. Effect of Germanium-Embedded Knee Sleeve on Osteoarthritis of the Knee. Orthop J Sports Med. 2019 Oct 25;7(10):2325967119879124. doi: 10.1177/2325967119879124. eCollection 2019 Oct. PMID 31696136
- [Background] Masiello F, Pati I, Veropalumbo E, Pupella S, Cruciani M, De Angelis V. Ultrasound-guided injection of platelet-rich plasma for tendinopathies: a systematic review and meta-analysis. Blood Transfus. 2023 Mar;21(2):119-136. doi: 10.2450/2022.0087-22. Epub 2022 Oct 17. PMID 36346880
- [Background] Lee SY, Kim W, Lim C, Chung SG. Treatment of Lateral Epicondylosis by Using Allogeneic Adipose-Derived Mesenchymal Stem Cells: A Pilot Study. Stem Cells. 2015 Oct;33(10):2995-3005. doi: 10.1002/stem.2110. Epub 2015 Aug 6. PMID 26202898
- [Background] Khoury M, Tabben M, Rolon AU, Levi L, Chamari K, D'Hooghe P. Promising improvement of chronic lateral elbow tendinopathy by using adipose derived mesenchymal stromal cells: a pilot study. J Exp Orthop. 2021 Jan 26;8(1):6. doi: 10.1186/s40634-020-00320-z. PMID 33501619
- [Background] Chen X, Jones IA, Park C, Vangsness CT Jr. The Efficacy of Platelet-Rich Plasma on Tendon and Ligament Healing: A Systematic Review and Meta-analysis With Bias Assessment. Am J Sports Med. 2018 Jul;46(8):2020-2032. doi: 10.1177/0363546517743746. Epub 2017 Dec 21. PMID 29268037
- [Background] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307
- [Background] Dejnek M, Moreira H, Placzkowska S, Barg E, Reichert P, Krolikowska A. Effectiveness of Lateral Elbow Tendinopathy Treatment Depends on the Content of Biologically Active Compounds in Autologous Platelet-Rich Plasma. J Clin Med. 2022 Jun 27;11(13):3687. doi: 10.3390/jcm11133687. PMID 35806972
- [Background] Kwapisz A, Prabhakar S, Compagnoni R, Sibilska A, Randelli P. Platelet-Rich Plasma for Elbow Pathologies: a Descriptive Review of Current Literature. Curr Rev Musculoskelet Med. 2018 Dec;11(4):598-606. doi: 10.1007/s12178-018-9520-1. PMID 30255288
- See also: Empowering Recovery: Surface Electromyography Shows how Incrediwear Helps Professional Athletes Recover — https://incrediwear.com/pages/research?srsltid=AfmBOooOWJNZ3dydamSCph_y8wrbqiv61n7MZ11508RRy9KeTgE3Am-0

DOCUMENTS (2):
  • Study Protocol (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT06846593/Prot_000.pdf
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT06846593/ICF_001.pdf